CLINICAL TRIAL: NCT01901432
Title: A Two-part Study Top Assess the Safety and Preliminary Efficacy of Givinostat in Patients With JAK2V617F Positive Polycythemia Vera
Brief Title: A Two-part Study to Assess the Safety and Preliminary Efficacy of Givinostat in Patients With Polycythemia Vera
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/12/2357/45; 2013-000860-27 (EudraCT Number)
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Polycythemia Vera
Keywords: chronic myeloproliferative neoplasms; Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis; Givinostat
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Givinostat (Experimental): In Part A patients will treated in dose levels at the following daily doses of Givinostat:
  * 50 mg b.i.d.,
  * 100 mg b.i.d.;
  * 150 mg b.i.d.,
  * 200 mg b.i.d.;
  * 150 mg t.i.d.;
  * 200 mg t.i.d.. Intermediate dose levels and, consequently, additionally dose levels may be used to establish the Maximum Tolerated Dose.
  In Part B patients will be treated at the Maximum Tolerated Dose established in Part A.
  The product will be supplied as hard gelatine capsules for oral administration at the strength of 50 mg, 75 mg and/or 100 mg each.
  Interventions: Drug: Givinostat

INTERVENTIONS:
Drug: Givinostat — In Part A patients will treated in dose levels at the following daily doses of Givinostat:
  * 50 mg b.i.d.,
  * 100 mg b.i.d.;
  * 150 mg b.i.d.,
  * 200 mg b.i.d.;
  * 150 mg t.i.d.;
  * 200 mg t.i.d.. Intermediate dose levels and, consequently, additionally dose levels may be used to establish the Maximum Tolerated Dose.
  In Part B patients will be treated at the Maximum Tolerated Dose established in Part A. The product will be supplied as hard gelatine capsules for oral administration at the strength of 50 mg, 75 mg and/or 100 mg each.
  Other Names: Givinostat (ITF2357)

SUMMARY:
This is a two-part, multicenter, open label, non-randomized, phase Ib/II study to assess the safety and tolerability, Maximum Tolerated Dose and preliminary efficacy of Givinostat in patients with JAK2V617F positive Polycythemia Vera. Part A is the dose finding part while Part B is assessing the preliminary efficacy. Patients will be enrolled either in Part A or Part B and transition from one part to the other is not allowed.

Eligible patients for this study will have a confirmed diagnosis of Polycythemia Vera according to the revised World Health Organization criteria. Only if the enrolment in Part A is slow (i.e. < 5 patients enrolled in 3 months), eligibility for this part of the study may be expanded to all patients with chronic myeloproliferative neoplasms.

Study therapy will be administered in 28 day cycles (4 weeks of treatment). Disease response will be evaluated according to the European LeukemiaNet criteria after 3 and 6 cycles (i.e. at weeks 12 and 24, respectively) of treatment with Givinostat for both parts of the study. All phlebotomies performed in the first 3 weeks of treatment will not be counted to assess the clinico-haematological response.

The study will last up to a maximum of 24 weeks of treatment. However, after completion of the trial, all patients achieving clinical benefit will be allowed to continue treatment with Givinostat (at the same dose and schedule) in a long-term study.

Safety will be monitored at each visit throughout the entire duration of the study. Treatment will be administered on an outpatient basis and patients will be followed regularly with physical and laboratory tests, as specified in the protocol; in case of hospitalization, the treatment will be continued or interrupted according to the Investigators' decision.

DETAILED DESCRIPTION:
This is a two-part, multicenter, open label, non-randomized, phase Ib/II study to assess the safety and tolerability, MTD and preliminary efficacy of Givinostat in patients with JAK2V617F positive PV.

Part A is the dose escalation portion of the study and, once the MTD has been established, Part B will commence where the preliminary efficacy of Givinostat in PV patients will be established. Patients will be enrolled either in Part A or Part B and transition from one part to the other is not allowed. Only PV patients from Part A assigned to the dose selected for Part B (MTD) may be counted towards the efficacy assessment in Part B.

Eligible patients for this study will have a confirmed diagnosis of PV according to the revised WHO criteria and the JAK2V617F positivity. Only if the enrolment in Part A is slow (i.e. < 5 patients enrolled in 3 months), eligibility for this part of the study may be expanded to all patients with cMPN.

After providing informed written consent before undertaking any protocol-related procedure, a unique patient identification code (i.e. patient screening ID which will be a combination of his/her site ID, study part ID and patient screening number, e.g. IT01-A01) will be assigned to each patient and it will identify the patient within his/her enrolment confirmation by Italfarmaco S.p.A. or its designee and never be reused in case of screening failure. After the enrolment confirmation and the assignation of the dose level before the first drug intake, a unique patient identification code (i.e. patient ID which will be a combination of patient screening number ID and dose level ID, e.g. IT01-A01-DL1) will be assigned to each patient and it will identify the patient throughout his/her participation in the study and never be reused in case of premature drop-out.

Study therapy will be administered in 28 day cycles. In fact, the "cycle" is defined as 4 weeks of treatment.

Disease response will be evaluated according to the clinico-haematological ELN criteria after 3 and 6 cycles (i.e. at weeks 12 and 24, respectively) of treatment with Givinostat for both parts of the study. All phlebotomies performed in the first 3 weeks of treatment will not be counted to assess the clinico-haematological response.

The study will last up to a maximum of 24 weeks of treatment. However, after completion of the trial, all patients achieving clinical benefit will be allowed to continue treatment with Givinostat (at the same dose and schedule) in a long-term study (Study N.: DSC/11/2357/44).

Safety will be monitored at each visit throughout the entire duration of the study. Treatment will be administered on an outpatient basis and patients will be followed regularly with physical and laboratory tests, as specified in the protocol; in case of hospitalization, the treatment will be continued or interrupted according to the Investigators' decision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to provide informed consent and be willing to sign an informed consent form;
2. Patients must have an age ≥18 years;
3. Patients must have a confirmed diagnosis of Polycythemia Vera according to the revised World Health Organization criteria;
4. Patients must have mutated Janus Kinase 2 (mutation V617F) positive disease;
5. Patients must have an active/not controlled disease defined as

   1. hematocrit ≥ 45% or hematocrit <45% in need of phlebotomy, and
   2. platelet count > 400 x109/L, and
   3. white blood cell count > 10 x109/L;
6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 in Part A, ECOG performance status ≤ 2 in Part B within 7 days of initiating study drug;
7. Female patient of childbearing potential has a negative serum or urine pregnancy test within 72 hours of the first dose of study therapy;
8. Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential;
9. Adequate and acceptable organ function within 7 days of initiating study drug;
10. Willingness and capability to comply with the requirements of the study.

Note that if the enrolment in Part A is slow (i.e. < 5 patients enrolled in 3 months), eligibility for this part of the study may be expanded to all patients with chronic myeloproliferative neoplasms. In this case, the inclusion criteria 5 will be modified as following only for Part A:

5. Patients must have an active/not controlled disease defined as:

1. Essential Thrombocythemia patients: Platelet count > 600 x109/L;
2. Myelofibrosis patients: no response according to European Myelofibrosis Network criteria.

Exclusion Criteria:

1. Active bacterial or mycotic infection requiring antimicrobial treatment;
2. Pregnancy or nursing;
3. A clinically significant corrected QT interval prolongation at baseline;
4. Use of concomitant medications known to prolong the corrected QT interval;
5. Clinically significant cardiovascular disease including:

   1. Uncontrolled hypertension despite medical treatment, myocardial infarction, unstable angina within 6 months from study start;
   2. New York Heart Association Grade II or greater congestive heart failure;
   3. History of any cardiac arrhythmia requiring medication (irrespective of its severity);
   4. A history of additional risk factors for torsade de pointes;
6. Known positivity for human immunodeficiency;
7. Known active hepatitis B virus and/or hepatitis C virus infection;
8. Platelet count < 100 x109/L within 14 days before enrolment;
9. Absolute neutrophil count < 1.2x109/L within 14 days before enrolment;
10. Serum creatinine > 2 times the upper limit of normal;
11. Total serum bilirubin > 1.5 times the upper limit of normal except in case of Gilbert's disease;
12. Serum aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 3 times the upper limit of normal;
13. History of other diseases (including active tumours), metabolic dysfunctions, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications;
14. Prior treatment with a Janus Kinase 2 or Histone Deacetylase inhibitor or participation in an interventional clinical trial for chronic myeloproliferative neoplasms;
15. Systemic treatment for chronic myeloproliferative neoplasms other than aspirin/cardio aspirin;
16. Hydroxyurea within 28 days before enrolment;
17. Interferon alpha within 14 days before enrolment;
18. Anagrelide within 7 days before enrolment;
19. Any other investigational drug or device within 28 days before enrolment;
20. Patient with known hypersensitivity to the components of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06-26 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bettica, MD, Study Director — Italfarmaco S.p.A.
Locations (25):
- France (4):
  - CHU Amiens - Hôpital Sud, Amiens
  - Hôpital Morvan - CHRU de Brest, Brest
  - Hopital Saint Vincent de Paul - GHICL Lille, Lille
  - Hôpital Saint-Louis (AP-HP), Centre Investigations Cliniques, Paris
- Germany (4):
  - Charite Research Organisation GmbH, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- Italy (12):
  - Azienda ospedaliero universitaria Consorziale Policlinico di Bari, Bari, BA
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, BG
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Florence, FI
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Istituto Tumori Giovanni Paolo II - IRCCS Ospedale Oncologico di Bari, Bari
  - Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico, Milan
  - Università degli Studi di Napoli Federico II, Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale Civile dello Spirito Santo, Pescara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera "Bianchi-Melacrino-Morelli", Reggio Calabria
  - Università Campus Bio-Medico di Roma, Rome
  - Ospedale San Bortolo di Vicenza, Vicenza
- Poland (2):
  - SP ZOZ Zespol Szpitali Miejskich w Chorzowie, Chorzów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
- United Kingdom (3):
  - Belfast City Hospital, Belfast
  - Royal London Hospital, London
  - Royal Cornwall Hospital, Truro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part, multisite, open-label, non-randomized study to assess givinostat in patients with JAK2^V617F positive Polycythemia Vera. Part A assessed safety and was the dose escalation portion of study, while Part B assessed preliminary efficacy. Patients were enrolled in 5 countries (France, Germany, Italy, Poland and the United Kingdom).
Pre-assignment Details: Patients were enrolled into either Part A or Part B, transition from 1 part to the other was not allowed. 48 patients were enrolled into the study overall: 12 patients in Part A to determine the maximum tolerated dose (MTD) and 36 patients in Part B.
Groups:
- Givinostat DL0 (50 mg b.i.d.) (Part A): In Part A, 3 patients were assigned to receive givinostat by oral administration at Dose Level 0 (DL0) (50 milligrams [mg] twice daily [b.i.d.]). Patients were treated for up to 6 cycles (28 days in each cycle).
  There were 3 DLs used during Part A; 50 mg b.i.d. (DL0) was the third DL to be administered.
- Givinostat DL1 (100 mg b.i.d.) (Part A): In Part A, 3 patients were assigned to receive givinostat by oral administration at DL1 (100 mg b.i.d.). Patients were treated for up to 6 cycles (28 days in each cycle).
  There were 3 DLs used during Part A; 100 mg b.i.d. (DL1) was the initial DL to be administered.
- Givinostat DL1 Expanded (100 mg b.i.d.) (Part A): Following initial assignment of 3 patients to DL1 in Part A, a further 3 patients were assigned to DL1 so this treatment group is referred to as "DL1 expanded" (patients received givinostat by oral administration at 100 mg b.i.d.). Patients were treated for up to 6 cycles (28 days in each cycle).
  There were 3 DLs used during Part A; 100 mg b.i.d. (DL1) was the initial DL to be administered.
- Givinostat DL6 (100 mg + 50 mg) (Part A): In Part A, 3 patients were assigned to receive givinostat by oral administration at DL6 (100 mg in the morning and 50 mg in the evening, i.e. 12 hours after). Patients were treated for up to 6 cycles in (28 days in each cycle).
  There were 3 DLs used during Part A; 100 mg + 50 mg (DL6) was the second DL to be administered.
- Givinostat at MTD (100 mg b.i.d.) (Part B): In Part B, patients were assigned to receive the starting dose of givinostat by oral administration at the MTD determined in Part A (i.e. 100 mg b.i.d.). Patients were treated for up to 6 cycles (28 days in each cycle). Based on evaluations performed as part of the visit procedures on Day 28 of each cycle up to Cycle 5 and/or in any necessary additional study visit, the givinostat dose was decreased if appropriate for any patients that met dose reduction criteria.
Period: Overall Study
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A) | Givinostat DL1 (100 mg b.i.d.) (Part A) | Givinostat DL1 Expanded (100 mg b.i.d.) (Part A) | Givinostat DL6 (100 mg + 50 mg) (Part A) | Givinostat at MTD (100 mg b.i.d.) (Part B)
Started | 3 | 3 | 3 | 3 | 36
Received Study Drug | 3 | 3 | 3 | 3 | 35
Completed | 3 | 2 | 1 | 3 | 27
Not Completed | 0 | 1 | 2 | 0 | 9
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Patient decision to stop study drug | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The overall baseline population consists of all enrolled patients in either Part A or Part B of the study.
Groups:
- Givinostat DL0 (50 mg b.i.d.) (Part A): In Part A, 3 patients were assigned to receive givinostat by oral administration at DL0 (50 mg twice daily [b.i.d.]). Patients were treated for up to 6 cycles (28 days in each cycle).
  There were 3 DLs used during Part A; 50 mg b.i.d. (DL0) was the third DL to be administered.
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A) | Givinostat DL1 (100 mg b.i.d.) (Part A) | Givinostat DL1 Expanded (100 mg b.i.d.) (Part A) | Givinostat DL6 (100 mg + 50 mg) (Part A) | Givinostat at MTD (100 mg b.i.d.) (Part B) | Total Title
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 36 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 2 | 28 | 35
  >=65 years | 1 | 1 | 2 | 1 | 8 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 11 | 16
  Male | 1 | 2 | 2 | 2 | 25 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 36 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Treatment-emergent Adverse Events (TEAEs) in Part A of the Study
Description: Evaluations were performed on the type, incidence and severity of TEAEs, graded according to Common Terminology Criteria for Adverse Events (CTCAE) v. 4.03, following administration of givinostat for up to 6 cycles of treatment in Part A. Grades 1 through 5 were as follows: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening or requiring hospitalisation; Grade 4: Life threatening consequences; Grade 5: Death related to AE. Results are reported as number of patients with TEAEs for each of the indicated categories. Definitions: drug-related TEAE / treatment-emergent serious adverse event (TESAE) corresponded to reasonable suspicion that the TEAE / TESAE was associated with the use of the study drug, according to investigator assessment; discontinuation refers to discontinuation from treatment.
Time Frame: 168 days (up to Cycle 6 Day 28 in Part A).
Population: The Safety (SAF) analysis set included all recruited patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Givinostat DL0 (50 mg b.i.d.) (Part A): In Part A, 3 patients were assigned to receive givinostat by oral administration at DL0 (50 mg b.i.d.). Patients were treated for up to 6 cycles (28 days in each cycle).
  There were 3 DLs used during Part A; 50 mg b.i.d. (DL0) was the third DL to be administered.
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A) | Givinostat DL1 (100 mg b.i.d.) (Part A) | Givinostat DL1 Expanded (100 mg b.i.d.) (Part A) | Givinostat DL6 (100 mg + 50 mg) (Part A)
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants
  TEAE | 3 | 3 | 3 | 3
  Drug-related TEAE | 1 | 3 | 3 | 1
  TESAE | 0 | 1 | 0 | 1
  Drug-related TESAE | 0 | 0 | 0 | 0
  Death due to any cause | 0 | 0 | 0 | 0
  Grade 3 TEAE | 0 | 2 | 1 | 1
  Grade 3 drug-related TEAE | 0 | 2 | 1 | 0
  Grade 4 TEAE | 0 | 0 | 1 | 0
  Grade 4 drug-related TEAE | 0 | 0 | 1 | 0
  Grade 5 TEAE | 0 | 0 | 0 | 0
  Discontinuation due to TEAE | 0 | 1 | 1 | 0
  Discontinuation due to drug-related TEAE | 0 | 1 | 1 | 0
  Discontinuation due to TESAE | 0 | 0 | 0 | 0
  Discontinuation due to drug-related TESAE | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) After 1 Cycle in Part A of the Study
Description: The MTD of givinostat was based only on Cycle 1 DLTs. A DLT was defined as the following drug-related toxicity:
  * Grade 4 hematological toxicity, or
  * Grade 3 febrile neutropenia, or
  * Grade ≥3 non-hematological toxicity (with the exception Grade 3 diarrhea without adequate supportive care lasting less than 3 days, and Grade 3 nausea or vomiting without adequate supportive care lasting less than 3 days), or
  * Any drug-related serious AE, or
  * Any toxicity clearly not related to disease progression or intercurrent illness requiring interruption of dosing for more than 3 days during first cycle.
  At end of Cycle 1, for the third patient in each DL, the safety of the 3 patients treated for 1 cycle was reviewed and it was decided if the dose should be escalated or not. Results are reported as the number of patients with DLT events for Cycle 1 in Part A.
Time Frame: 28 days (up to Cycle 1 Day 28 in Part A).
Population: The MTD analysis set included all patients who experienced a DLT in Cycle 1 of Part A, or received ≥90% of study drug doses in Cycle 1 of Part A.
Measure: Number; unit: participants
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A) | Givinostat DL1 (100 mg b.i.d.) (Part A) | Givinostat DL1 Expanded (100 mg b.i.d.) (Part A) | Givinostat DL6 (100 mg + 50 mg) (Part A)
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Patients Experiencing TEAEs After 3 Cycles in Part B of the Study
Description: Evaluations were performed on the type, incidence and severity of TEAEs, graded according to CTCAE v. 4.03, following administration of givinostat at the MTD for up to 3 cycles of treatment in Part B. Grades 1 through 5 were as follows: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening or requiring hospitalisation; Grade 4: Life threatening consequences; Grade 5: Death related to AE. Results are reported as number of patients with TEAEs for each of the indicated categories. Definitions: drug-related TEAE / TESAE corresponded to reasonable suspicion that the TEAE / TESAE was associated with the use of the study drug, according to investigator assessment; discontinuation refers to discontinuation from treatment.
Time Frame: 84 days (up to Cycle 3 Day 28 in Part B).
Population: The SAF analysis set included all recruited patients who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Givinostat at MTD (100 mg b.i.d.) (Part B)
Number analyzed (Participants) | 35
Participants
  TEAE | 35
  Drug-related TEAE | 33
  TESAE | 2
  Drug-related TESAE | 1
  Death due to any cause | 0
  Grade 3 TEAE | 10
  Grade 3 drug-related TEAE | 7
  Grade 4 TEAE | 0
  Grade 4 drug-related TEAE | 0
  Grade 5 TEAE | 0
  Discontinuation due to TEAE | 2
  Discontinuation due to drug-related TEAE | 2
  Discontinuation due to TESAE | 0
  Discontinuation due to drug-related TESAE | 0

4. Primary Outcome: Overall Response Rate (ORR) (i.e. Complete Response [CR] and Partial Response [PR]) After 3 Cycles in Part B of the Study
Description: ORR, CR and PR following administration of givinostat at MTD for 3 cycles in Part B, reported as percentage of patients with a response. Response was evaluated according to the clinico-hematological European LeukemiaNet (ELN) response criteria. If Investigator's clinical response assessment (taking into account the overall medical judgment of the specific patient's case) was not in agreement with exact application of the ELN response criteria, the Investigator's assessment superseded the mathematical application of these criteria and was used for analysis.
  CR defined as:
  1. Hematocrit (HCT) <45% without phlebotomy, and
  2. Platelets ≤400 x10^9/litre (L), and
  3. White Blood Cell count ≤10 x10^9/L, and
  4. Normal spleen size, and
  5. No disease-related systemic symptoms (i.e. pruritus, headache, microvascular disturbances).
  PR defined as: Patients not fulfilling CR and
  1. HCT <45% without phlebotomy, or
  2. Response in ≥3 other criteria.
Time Frame: 84 days (up to cycle 3 Day 28 in Part B).
Population: The Intent-to-Treat (ITT) analysis set included all recruited patients who received ≥1 dose of study drug and from whom ≥1 post-baseline efficacy measurement was obtained.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Givinostat at MTD (100 mg b.i.d.) (Part B)
Number analyzed (Participants) | 31
percentage of participants
  ORR (CR + PR) | 80.6 [62.53 to 92.55]
  CR | 9.7 [2.04 to 25.75]
  PR | 71.0 [51.96 to 85.78]

5. Secondary Outcome: ORR After 3 Cycles and After 6 Cycles in Part A of the Study
Description: ORR following administration of givinostat after 3 cycles and after 6 cycles in Part A, reported as percentage of patients with a response. Response was evaluated according to the clinico-hematological ELN response criteria. If Investigator's clinical response assessment (taking into account the overall medical judgment of the specific patient's case) was not in agreement with exact application of the ELN response criteria, the Investigator's assessment superseded the mathematical application of these criteria and was used for analysis. Analysis performed using the dataset for all Part A patients combined.
Time Frame: 84 and 168 days (up to Cycle 3 Day 28 and Cycle 6 Day 28 in Part A).
Population: The ITT analysis set included all recruited patients who received ≥1 dose of study drug and from whom ≥1 post-baseline efficacy measurement was obtained.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Givinostat Total (Part A): This dataset comprised all patients in the ITT analysis set who received givinostat in Part A of the study. It represents the 4 Part A treatment arms and includes patients who received givinostat at DL0 (50 mg b.i.d.), DL1 (100 mg b.i.d. [i.e. including DL1 expanded] and DL6 (100 mg + 50 mg) in Part A.
Arm/Group | Givinostat Total (Part A)
Number analyzed (Participants) | 11
percentage of participants
  Cycle 3 Day 28 | 72.7 [39.03 to 93.98]
  Cycle 6 Day 28 | 72.7 [39.03 to 93.98]

6. Secondary Outcome: ORR After 6 Cycles in Part B of the Study
Description: ORR following administration of givinostat at the MTD for 6 cycles in Part B, reported as percentage of patients with a response. Response was evaluated according to the clinico-hematological ELN response criteria. If Investigator's clinical response assessment (taking into account the overall medical judgment of the specific patient's case) was not in agreement with exact application of the ELN response criteria, the Investigator's assessment superseded the mathematical application of these criteria and was used for analysis.
Time Frame: 168 days (up to Cycle 6 Day 28 in Part B).
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Givinostat at MTD (100 mg b.i.d.) (Part B)
Number analyzed (Participants) | 31
percentage of participants | 80.6 [62.53 to 92.55]

7. Secondary Outcome: Number of Patients Experiencing TEAEs After 6 Cycles in Part B of the Study
Description: Evaluations were performed on the type, incidence and severity of TEAEs, graded according to CTCAE v. 4.03, following administration of givinostat at the MTD for up to 6 cycles of treatment in Part B. Grades 1 through 5 were as follows: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening or requiring hospitalisation; Grade 4: Life threatening consequences; Grade 5: Death related to AE. Results are reported as number of patients with TEAEs for each of the indicated categories. Definitions: drug-related TEAE / TESAE corresponded to reasonable suspicion that the TEAE / TESAE was associated with the use of the study drug, according to investigator assessment; discontinuation refers to discontinuation from treatment. Results are reported as number of patients with TEAEs for each of the indicated categories.
Time Frame: 168 days (up to Cycle 6 Day 28 in Part B).
Population: The SAF analysis set included all recruited patients who received ≥1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Givinostat at MTD (100 mg b.i.d.) (Part B)
Number analyzed (Participants) | 35
participants
  TEAE | 35
  Drug-related TEAE | 33
  TESAE | 2
  Drug-related TESAE | 1
  Death due to any cause | 0
  Grade 3 TEAE | 12
  Grade 3 drug-related TEAE | 10
  Grade 4 TEAE | 0
  Grade 4 drug-related TEAE | 0
  Grade 5 TEAE | 0
  Discontinuation due to TEAE | 2
  Discontinuation due to drug-related TEAE | 2
  Discontinuation due to TESAE | 0
  Discontinuation due to drug-related TESAE | 0

8. Secondary Outcome: Assessment of Maximum Plasma Concentration (Cmax) of Givinostat and Metabolites (ITF2374 and ITF2375) in Part A of the Study
Description: Pharmacokinetic (PK) evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of Cmax following administration of givinostat for 1 cycle in Part A. PK calculations were performed by standard non-compartmental analysis. Results are reported for Cycle 1 Day 1 and Cycle 1 Day 28.
  Note: concentration data for ITF2374 (Cycle 1 Day 1 and Cycle 1 Day 28) and for ITF2375 (Cycle 1 Day 1) in the DL0 dose group of Part A were not available for PK analysis.
Time Frame: Blood samples were collected in Part A on Cycle 1 Day 1: pre-dose and 2, 3 and 8 hours post-dose; and on Cycle 1 Day 28: pre-dose and 1, 2, 4 and 8 hours post-dose.
Population: The PK analysis set included all SAF patients with at least 1 PK assessment. Only patients with data available for analysis at each time point are presented.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Groups:
- Givinostat DL0 (50 mg b.i.d.) (Part A PK Analysis Set): This dataset was used for PK analysis and included the patients who received givinostat at DL0 (50 mg b.i.d.) in Part A of the study and for whom PK data was available for analysis.
- Givinostat DL1 (100 mg b.i.d.) (Part A PK Analysis Set): This dataset was used for PK analysis and included the patients who received givinostat at DL1 (100 mg b.i.d. [i.e. including DL1 expanded]) in Part A of the study and for whom PK data was available for analysis.
- Givinostat DL6 (100 mg + 50 mg) (Part A PK Analysis Set): This dataset was used for PK analysis and included the patients who received givinostat at DL6 (100 mg in the morning and 50 mg in the evening) in Part A of the study and for whom PK data was available for analysis.
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL1 (100 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL6 (100 mg + 50 mg) (Part A PK Analysis Set)
Number analyzed (Participants) | 3 | 6 | 3
nanograms per millilitre (ng/mL)
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 3
  Givinostat Cycle 1 Day 1 | 60.2 (43.1) | 54.3 (17.2) | 82.5 (24.4)
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 0 | 5 | 3
  ITF2374 Cycle 1 Day 1 |  | 3.74 (4.09) | 5.69 (2.87)
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 0 | 5 | 2
  ITF2375 Cycle 1 Day 1 |  | 68.6 (21.2) | 101 (24.5)
  Givinostat Cycle 1 Day 28: number analyzed (Participants) | 3 | 4 | 3
  Givinostat Cycle 1 Day 28 | 22.4 (8.92) | 73.3 (31.9) | 290 (330)
  ITF2374 Cycle 1 Day 28: number analyzed (Participants) | 0 | 4 | 3
  ITF2374 Cycle 1 Day 28 |  | 19.7 (7.24) | 31.3 (4.95)
  ITF2375 Cycle 1 Day 28: number analyzed (Participants) | 2 | 4 | 3
  ITF2375 Cycle 1 Day 28 | 110 (22.8) | 259 (75.9) | 376 (215)

9. Secondary Outcome: Assessment of Time to Maximum Plasma Concentration (Tmax) of Givinostat and Metabolites (ITF2374 and ITF2375) in Part A of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of Tmax following administration of givinostat for 1 cycle in Part A. PK calculations were performed by standard non-compartmental analysis. Results are reported for Cycle 1 Day 1 and Cycle 1 Day 28.
  Note: concentration data for ITF2374 (Cycle 1 Day 1 and Cycle 1 Day 28) and for ITF2375 (Cycle 1 Day 1) in the DL0 dose group of Part A were not available for PK analysis.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL1 (100 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL6 (100 mg + 50 mg) (Part A PK Analysis Set)
Number analyzed (Participants) | 3 | 6 | 3
hours
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 3
  Givinostat Cycle 1 Day 1 | 2.00 [1.92 to 3.00] | 2.00 [2.00 to 2.00] | 3.00 [2.00 to 3.00]
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 0 | 4 | 3
  ITF2374 Cycle 1 Day 1 |  | 8.00 [8.00 to 8.00] | 8.00 [3.00 to 8.00]
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 0 | 5 | 2
  ITF2375 Cycle 1 Day 1 |  | 3.00 [2.00 to 3.00] | 2.50 [2.00 to 3.00]
  Givinostat Cycle 1 Day 28: number analyzed (Participants) | 3 | 4 | 3
  Givinostat Cycle 1 Day 28 | 3.90 [3.83 to 4.00] | 1.50 [1.00 to 3.98] | 2.05 [1.05 to 4.00]
  ITF2374 Cycle 1 Day 28: number analyzed (Participants) | 0 | 4 | 3
  ITF2374 Cycle 1 Day 28 |  | 8.00 [0.00 to 8.00] | 2.00 [1.05 to 4.05]
  ITF2375 Cycle 1 Day 28: number analyzed (Participants) | 2 | 4 | 3
  ITF2375 Cycle 1 Day 28 | 2.00 [2.00 to 2.00] | 1.99 [1.00 to 3.98] | 4.00 [0.00 to 4.05]

10. Secondary Outcome: Assessment of Time of the Last Detectable Concentration (Tlast) of Givinostat and Metabolites (ITF2374 and ITF2375) in Part A of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of Tlast following administration of givinostat for 1 cycle in Part A. PK calculations were performed by standard non-compartmental analysis. Results are reported for Cycle 1 Day 1 and Cycle 1 Day 28.
  Note: concentration data for ITF2374 (Cycle 1 Day 1 and Cycle 1 Day 28) and for ITF2375 (Cycle 1 Day 1) in the DL0 dose group of Part A were not available for PK analysis.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL1 (100 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL6 (100 mg + 50 mg) (Part A PK Analysis Set)
Number analyzed (Participants) | 3 | 6 | 3
hours
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 3
  Givinostat Cycle 1 Day 1 | 7.97 (0.0462) | 8.00 (0.00) | 8.00 (0.00)
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 0 | 4 | 3
  ITF2374 Cycle 1 Day 1 |  | 8.00 (0.00) | 8.00 (0.00)
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 0 | 5 | 2
  ITF2375 Cycle 1 Day 1 |  | 8.00 (0.00) | 8.00 (0.00)
  Givinostat Cycle 1 Day 28: number analyzed (Participants) | 3 | 4 | 3
  Givinostat Cycle 1 Day 28 | 8.05 (0.249) | 7.00 (2.01) | 8.02 (0.0252)
  ITF2374 Cycle 1 Day 28: number analyzed (Participants) | 0 | 4 | 3
  ITF2374 Cycle 1 Day 28 |  | 7.00 (2.01) | 8.02 (0.0252)
  ITF2375 Cycle 1 Day 28: number analyzed (Participants) | 2 | 4 | 3
  ITF2375 Cycle 1 Day 28 | 3.00 (1.41) | 7.00 (2.01) | 6.70 (2.30)

11. Secondary Outcome: Assessment of Area Under Plasma Concentration Versus the Time Curve up to the Last Detectable Concentration (AUClast) of Givinostat and Metabolites (ITF2374 and ITF2375) in Part A of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of AUClast following administration of givinostat for 1 cycle in Part A. PK calculations were performed by standard non-compartmental analysis and AUClast was calculated using the linear trapezoidal rule. Results are reported for Cycle 1 Day 1 and Cycle 1 Day 28.
  Note: concentration data for ITF2374 (Cycle 1 Day 1 and Cycle 1 Day 28) and for ITF2375 (Cycle 1 Day 1) in the DL0 dose group of Part A were not available for PK analysis.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL1 (100 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL6 (100 mg + 50 mg) (Part A PK Analysis Set)
Number analyzed (Participants) | 3 | 6 | 3
ng*h/mL
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 3
  Givinostat Cycle 1 Day 1 | 208 (136) | 238 (55.6) | 429 (109)
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 0 | 5 | 3
  ITF2374 Cycle 1 Day 1 |  | 14.4 (19.0) | 29.6 (9.64)
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 0 | 5 | 2
  ITF2375 Cycle 1 Day 1 |  | 416 (153) | 611 (146)
  Givinostat Cycle 1 Day 28: number analyzed (Participants) | 3 | 4 | 3
  Givinostat Cycle 1 Day 28 | 132 (45.1) | 359 (203) | 1100 (1050)
  ITF2374 Cycle 1 Day 28: number analyzed (Participants) | 0 | 4 | 3
  ITF2374 Cycle 1 Day 28 |  | 102 (11.7) | 158 (42.6)
  ITF2375 Cycle 1 Day 28: number analyzed (Participants) | 2 | 4 | 3
  ITF2375 Cycle 1 Day 28 | 263 (192) | 1390 (675) | 1780 (1190)

12. Secondary Outcome: Assessment of Area Under Plasma Concentration Versus the Time Curve in the Dosing Interval (0-12 Hours) (AUC0-12) of Givinostat and Metabolites (ITF2374 and ITF2375) in Part A of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of AUC0-12 following administration of givinostat for 1 cycle in Part A. PK calculations were performed by standard non-compartmental analysis and AUC0-12 was calculated using the linear trapezoidal rule. Results are reported for Cycle 1 Day 1 and Cycle 1 Day 28.
  Note:concentration data for ITF2374 (Cycle 1 Day 1 and Cycle 1 Day 28) across all dose groups and for ITF2375 (Cycle 1 Day 1) in the DL0 dose group of Part A were not available for PK analysis.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL1 (100 mg b.i.d.) (Part A PK Analysis Set) | Givinostat DL6 (100 mg + 50 mg) (Part A PK Analysis Set)
Number analyzed (Participants) | 3 | 6 | 3
ng*h/mL
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 3 | 5 | 3
  Givinostat Cycle 1 Day 1 | 235 (146) | 289 (68.9) | 508 (107)
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 0 | 5 | 2
  ITF2375 Cycle 1 Day 1 |  | 598 (259) | 870 (182)
  Givinostat Cycle 1 Day 28: number analyzed (Participants) | 3 | 3 | 3
  Givinostat Cycle 1 Day 28 | 161 (51.8) | 533 (223) | 1180 (1050)
  ITF2374 Cycle 1 Day 28: number analyzed (Participants) | 0 | 0 | 0
  ITF2375 Cycle 1 Day 28: number analyzed (Participants) | 1 | 3 | 3
  ITF2375 Cycle 1 Day 28 | 863 (NA) — NA=Not available. Only 1 patient analyzed for this parameter so standard deviation value is not applicable. | 2020 (1000) | 2340 (970)

13. Secondary Outcome: Assessment of Cmax of Givinostat and Metabolites (ITF2374 and ITF2375) in Part B of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of Cmax following administration of givinostat for 2 cycles in Part B. PK calculations were performed by standard non-compartmental analysis. Following definition of the MTD in Part A, during Part B Cycle 1, givinostat was administered at 100 mg b.i.d. and during Part B Cycle 2 was administered at 100 mg, 75 mg and 50 mg b.i.d. (since dose reductions due to TEAEs were allowed from Cycle 2 onwards, as per protocol). Results are reported for Cycle 1 Day 1 and Cycle 2 Day 28 for the doses administered during Part B.
  Note: PK evaluation for the givinostat 75 mg and 50 mg b.i.d. dose groups for Cycle 1 Day 1 was not applicable (since all received givinostat 100 mg b.i.d.). Additionally, concentration data for ITF2375 (Cycle 1 Day 28) in the 50 mg b.i.d. dose group was not available for PK analysis.
Time Frame: Blood samples were collected in Part B on Cycle 1 Day 1: pre-dose and 2, 3 and 8 hours post-dose; and on Cycle 2 Day 28: pre-dose and 1, 2, 4 and 8 hours post-dose.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Givinostat 100 mg b.i.d. (Part B PK Analysis Set): This dataset was used for PK analysis and included patients who received givinostat at the MTD (100 mg b.i.d.) in Part B of the study and for whom PK data was available for analysis. This dataset was used for PK analysis after Cycle 1 Day 1 (34 patients) and after Cycle 2 Day 28 (17 patients remaining at this dose).
- Givinostat 75 mg b.i.d. (Part B PK Analysis Set): This dataset was used for PK analysis and included patients who received givinostat at the reduced dose of 75 mg b.i.d. in Part B of the study and for whom PK data was available for analysis. This dataset only applied for PK analysis from Cycle 2 onwards (i.e. Cycle 2 Day 28).
- Givinostat 50 mg b.i.d. (Part B PK Analysis Set): This dataset was used for PK analysis and included patients who received givinostat at the reduced dose of 50 mg b.i.d. in Part B of the study and for whom PK data was available for analysis. This dataset only applied for PK analysis from Cycle 2 onwards (i.e. Cycle 2 Day 28).
Arm/Group | Givinostat 100 mg b.i.d. (Part B PK Analysis Set) | Givinostat 75 mg b.i.d. (Part B PK Analysis Set) | Givinostat 50 mg b.i.d. (Part B PK Analysis Set)
Number analyzed (Participants) | 34 | 12 | 2
ng/mL
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  Givinostat Cycle 1 Day 1 | 71.5 (34.4) |  |
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  ITF2374 Cycle 1 Day 1 | 7.85 (4.89) |  |
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 29 | 0 | 0
  ITF2375 Cycle 1 Day 1 | 161 (72.9) |  |
  Givinostat Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  Givinostat Cycle 2 Day 28 | 90.8 (33.5) | 64.0 (22.6) | 62.6 (21.8)
  ITF2374 Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  ITF2374 Cycle 2 Day 28 | 32.3 (21.0) | 22.6 (11.2) | 21.4 (0.424)
  ITF2375 Cycle 2 Day 28: number analyzed (Participants) | 16 | 9 | 0
  ITF2375 Cycle 2 Day 28 | 320 (238) | 203 (78.7) |

14. Secondary Outcome: Assessment of Tmax of Givinostat and Metabolites (ITF2374 and ITF2375) in Part B of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of Tmax following administration of givinostat for 2 cycles in Part B. PK calculations were performed by standard non-compartmental analysis. Following definition of the MTD in Part A, during Part B Cycle 1, givinostat was administered at 100 mg b.i.d. and during Part B Cycle 2 was administered at 100 mg, 75 mg and 50 mg b.i.d. (since dose reductions due to TEAEs were allowed from Cycle 2 onwards, as per protocol). Results are reported for Cycle 1 Day 1 and Cycle 2 Day 28 for the doses administered during Part B.
  Note: PK evaluation for the givinostat 75 mg and 50 mg b.i.d. dose groups for Cycle 1 Day 1 was not applicable (since all received givinostat 100 mg b.i.d.). Additionally, concentration data for ITF2375 (Cycle 1 Day 28) in the 50 mg b.i.d. dose group was not available for PK analysis.
Time Frame: as for outcome 13
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Givinostat 100 mg b.i.d. (Part B PK Analysis Set) | Givinostat 75 mg b.i.d. (Part B PK Analysis Set) | Givinostat 50 mg b.i.d. (Part B PK Analysis Set)
Number analyzed (Participants) | 34 | 12 | 2
hours
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  Givinostat Cycle 1 Day 1 | 2.00 [0.00 to 8.00] |  |
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  ITF2374 Cycle 1 Day 1 | 8.00 [2.08 to 8.17] |  |
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 29 | 0 | 0
  ITF2375 Cycle 1 Day 1 | 3.00 [1.83 to 8.00] |  |
  Givinostat Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  Givinostat Cycle 2 Day 28 | 2.00 [0.00 to 4.07] | 2.00 [1.00 to 8.00] | 0.985 [0.00 to 1.97]
  ITF2374 Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  ITF2374 Cycle 2 Day 28 | 4.00 [0.00 to 8.00] | 3.04 [1.00 to 8.00] | 5.99 [3.97 to 8.00]
  ITF2375 Cycle 2 Day 28: number analyzed (Participants) | 16 | 9 | 0
  ITF2375 Cycle 2 Day 28 | 2.00 [0.00 to 4.00] | 2.00 [1.00 to 8.00] |

15. Secondary Outcome: Assessment of Tlast of Givinostat and Metabolites (ITF2374 and ITF2375) in Part B of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of Tlast following administration of givinostat for 2 cycles in Part B. PK calculations were performed by standard non-compartmental analysis. Following definition of the MTD in Part A, during Part B Cycle 1, givinostat was administered at 100 mg b.i.d. and during Part B Cycle 2 was administered at 100 mg, 75 mg and 50 mg b.i.d. (since dose reductions due to TEAEs were allowed from Cycle 2 onwards, as per protocol). Results are reported for Cycle 1 Day 1 and Cycle 2 Day 28 for the doses administered during Part B.
  Note: PK evaluation for the givinostat 75 mg and 50 mg b.i.d. dose groups for Cycle 1 Day 1 was not applicable (since all received givinostat 100 mg b.i.d.). Additionally, concentration data for ITF2375 (Cycle 1 Day 28) in the 50 mg b.i.d. dose group was not available for PK analysis.
Time Frame: as for outcome 13
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Givinostat 100 mg b.i.d. (Part B PK Analysis Set) | Givinostat 75 mg b.i.d. (Part B PK Analysis Set) | Givinostat 50 mg b.i.d. (Part B PK Analysis Set)
Number analyzed (Participants) | 34 | 12 | 2
hours
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  Givinostat Cycle 1 Day 1 | 7.42 (1.61) |  |
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  ITF2374 Cycle 1 Day 1 | 7.42 (1.61) |  |
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 29 | 0 | 0
  ITF2375 Cycle 1 Day 1 | 8.00 (0.0505) |  |
  Givinostat Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  Givinostat Cycle 2 Day 28 | 8.00 (0.0340) | 7.98 (0.0753) | 7.99 (0.0212)
  ITF2374 Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  ITF2374 Cycle 2 Day 28 | 8.00 (0.0340) | 7.98 (0.0753) | 7.99 (0.0212)
  ITF2375 Cycle 2 Day 28: number analyzed (Participants) | 16 | 9 | 0
  ITF2375 Cycle 2 Day 28 | 7.75 (1.00) | 8.00 (0.00) |

16. Secondary Outcome: Assessment of AUClast of Givinostat and Metabolites (ITF2374 and ITF2375) in Part B of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of AUClast following administration of givinostat for 2 cycles in Part B. PK calculations were performed by standard non-compartmental analysis and AUClast was calculated using the linear trapezoidal rule. Following definition of the MTD in Part A, during Part B Cycle 1, givinostat was administered at 100 mg b.i.d. and during Part B Cycle 2 was administered at 100 mg, 75 mg and 50 mg b.i.d. (since dose reductions due to TEAEs were allowed from Cycle 2 onwards, as per protocol). Results are reported for Cycle 1 Day 1 and Cycle 2 Day 28 for the for the doses administered during Part B.
  Note: PK evaluation for the givinostat 75 mg and 50 mg b.i.d. dose groups for Cycle 1 Day 1 was not applicable (since all received givinostat 100 mg b.i.d.). Additionally, concentration data for ITF2375 (Cycle 1 Day 28) in the 50 mg b.i.d. dose group was not available for PK analysis.
Time Frame: as for outcome 13
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Givinostat 100 mg b.i.d. (Part B PK Analysis Set) | Givinostat 75 mg b.i.d. (Part B PK Analysis Set) | Givinostat 50 mg b.i.d. (Part B PK Analysis Set)
Number analyzed (Participants) | 34 | 12 | 2
ng*h/mL
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  Givinostat Cycle 1 Day 1 | 289 (130) |  |
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 34 | 0 | 0
  ITF2374 Cycle 1 Day 1 | 28.5 (14.0) |  |
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 29 | 0 | 0
  ITF2375 Cycle 1 Day 1 | 888 (439) |  |
  Givinostat Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  Givinostat Cycle 2 Day 28 | 459 (145) | 323 (107) | 269 (78.5)
  ITF2374 Cycle 2 Day 28: number analyzed (Participants) | 17 | 12 | 2
  ITF2374 Cycle 2 Day 28 | 216 (127) | 161 (83.5) | 145 (20.9)
  ITF2375 Cycle 2 Day 28: number analyzed (Participants) | 16 | 9 | 0
  ITF2375 Cycle 2 Day 28 | 1830 (1660) | 1210 (585) |

17. Secondary Outcome: Assessment of AUC0-12 of Givinostat and Metabolites (ITF2374 and ITF2375) in Part B of the Study
Description: PK evaluation of givinostat and metabolites (ITF2374 and ITF2375) by assessment of AUC0-12 following administration of givinostat for 2 cycles in Part B. PK calculations were performed by standard non-compartmental analysis and AUClast was calculated using the linear trapezoidal rule. Following definition of the MTD in Part A, during Part B Cycle 1, givinostat was administered at 100 mg b.i.d. and during Part B Cycle 2 was administered at 100 mg, 75 mg and 50 mg b.i.d. (since dose reductions due to TEAEs were allowed from Cycle 2 onwards, as per protocol). Results are reported for Cycle 1 Day 1 and Cycle 2 Day 28 for the doses administered during Part B.
  Note: PK evaluation for the givinostat 75 mg and 50 mg b.i.d. dose groups for Cycle 1 Day 1 was not applicable (since all received givinostat 100 mg b.i.d.). Additionally, concentration data for ITF2374 (Cycle 1 Day 28) across all dose groups and for ITF2375 in the 50 mg b.i.d. dose group was not available for PK analysis.
Time Frame: as for outcome 13
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Givinostat 100 mg b.i.d. (Part B PK Analysis Set) | Givinostat 75 mg b.i.d. (Part B PK Analysis Set) | Givinostat 50 mg b.i.d. (Part B PK Analysis Set)
Number analyzed (Participants) | 34 | 12 | 2
ng*h/mL
  Givinostat Cycle 1 Day 1: number analyzed (Participants) | 29 | 0 | 0
  Givinostat Cycle 1 Day 1 | 372 (137) |  |
  ITF2374 Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0
  ITF2375 Cycle 1 Day 1: number analyzed (Participants) | 22 | 0 | 0
  ITF2375 Cycle 1 Day 1 | 1080 (619) |  |
  Givinostat Cycle 2 Day 28: number analyzed (Participants) | 17 | 11 | 2
  Givinostat Cycle 2 Day 28 | 561 (176) | 410 (129) | 326 (54.0)
  ITF2374 Cycle 2 Day 28: number analyzed (Participants) | 0 | 0 | 0
  ITF2375 Cycle 2 Day 28: number analyzed (Participants) | 14 | 7 | 0
  ITF2375 Cycle 2 Day 28 | 2460 (2450) | 1460 (608) |

ADVERSE EVENTS:
Time Frame: 168 days for Part A and 168 days for Part B (Cycle 1 through Cycle 6 for each phase of study; each cycle 28 days).
Description: TEAEs are reported for Part A and Part B and include events with an onset on or after the first administration of study drug until the end of study visit (or 7 days after the last drug intake for any patient permanently discontinuing study treatment).
Arm/Group | Givinostat DL0 (50 mg b.i.d.) (Part A) | Givinostat DL1 (100 mg b.i.d.) (Part A) | Givinostat DL1 Expanded (100 mg b.i.d.) (Part A) | Givinostat DL6 (100 mg + 50 mg) (Part A) | Givinostat at MTD (100 mg b.i.d.) (Part B)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 1/3 | 2/35
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Givinostat DL0 (50 mg b.i.d.) (Part A) (N=3) | Givinostat DL1 (100 mg b.i.d.) (Part A) (N=3) | Givinostat DL1 Expanded (100 mg b.i.d.) (Part A) (N=3) | Givinostat DL6 (100 mg + 50 mg) (Part A) (N=3) | Givinostat at MTD (100 mg b.i.d.) (Part B) (N=35)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Givinostat DL0 (50 mg b.i.d.) (Part A) (N=3) | Givinostat DL1 (100 mg b.i.d.) (Part A) (N=3) | Givinostat DL1 Expanded (100 mg b.i.d.) (Part A) (N=3) | Givinostat DL6 (100 mg + 50 mg) (Part A) (N=3) | Givinostat at MTD (100 mg b.i.d.) (Part B) (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (14)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 16 (22)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 8 (9)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 2 (4) | 2 (3) | 2 (5) | 20 (39)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 5 (5)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (13)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 10 (22)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 14 (21)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 3 (3)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Erythromelalgia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT01901432/SAP_000.pdf
  • Study Protocol (2015-07-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT01901432/Prot_001.pdf